CLINICAL TRIAL: NCT05099016
Title: Taking Action to Better Manage Cannabis Use Among Young Adults: Preliminary Evaluation of a Digital Tailored Prevention Tool With a Pilot Randomized Control Trial
Brief Title: Joint Effort Study
Acronym: JointEffort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21.196
Record Dates: First submitted 2021-08-31; First posted 2021-10-29 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2021-08

CONDITIONS: Cannabis Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint Effort (mobile application) (Experimental): The Joint Effort mobile application aims to support young adults into taking action on their cannabis use. Based on the Theory of Planned Behaviour, the content focuses on intention, attitude and perceived behavioral control. Various intervention methods and strategies are used to address these determinants (e.g., personalized feedback, persuasive communication, self-observation and activation of intention). The objectives includes: to allow the individual to become aware (or more aware) of their cannabis use, to support the individual's decision-making process of taking action on their cannabis use, to guide and support the establishment and sustainability of an action plan. An optional logbook-type feature (weekly journal of cannabis use) allows personalized monitoring and data collection throughout the course of the intervention.
  Interventions: Other: Joint Effort
- Brief normative feedback and standard information (Active Comparator): The comparator is composed of a a brief normative feedback regarding last month frequency of cannabis use and basic reliable non personalized information on lower-risk cannabis use (official public websites).
  Interventions: Other: Brief normative feedback and standard information

INTERVENTIONS:
Other: Joint Effort — The Joint Effort intervention is available in the form of an iPhone mobile application (running on iOS 13 and 14) in French language. It aims to support young adults in school who have used cannabis in the past month into taking action on their cannabis use.
  Arms: Joint Effort (mobile application)
Other: Brief normative feedback and standard information — The brief normative feedback is based on the frequency of cannabis use use. Participants will also be offered basic reliable non personalized information on lower-risk cannabis use in the form of official public websites.
  Arms: Brief normative feedback and standard information

SUMMARY:
This pilot randomized controlled trial (RCT) will be conducted to evaluate the acceptability and feasibility of a digital tailored prevention tool (i.e., the Joint Effort mobile application) aimed at supporting university-level students into taking action on their cannabis use. The two main objectives of the proposed study are:

1. To assess the acceptability of the Joint Effort mobile application in terms of uptake, engagement and intervention appreciation.
2. To document the feasibility of the study processes in terms of online recruitment rate, adherence to online data collection methods, and attrition rate.

ELIGIBILITY:
Inclusion Criteria:

* active cannabis user (i.e., having used cannabis at least once in the past month)
* able to understand French
* own an iPhone (running on iOS 13 or higher).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Uptake of the developed mobile application (acceptability) | 6 months
  Uptake is defined as the act of downloading and installing the mobile application (Szinay, Jones, Chadborn, Brown, & Naughton, 2020). The uptake rate will measure the proportion of participants randomized to the EG group that downloaded the mobile application (via the Apple iOS App Store) versus those who did not do it.
Subjective engagement with the developed mobile application (acceptability) | 4-weeks post baseline
  Subjective engagement (self-reported) will be measured by using the validated French version (Fontaine et al., 2020) of the User Engagement Scale - Short Form (UES-SF)(O'Brien et al., 2018). This 12-item instrument serves to measure four dimensions of engagement: 1) aesthetic appeal; 2) focused attention; 3) perceived usability; and 4) reward factor. Possible answers range from strongly disagree (+1) to strongly agree (+5). The possible total score ranges between 12 and 60. The score for each item will be interpreted and the scores for each dimensions will be compared to indicate which are rated more highly than other.
Objective engagement with the developed mobile application (acceptability) | 6 months
  Objective engagement (ie. number of screens viewed by participants) will be assessed. This data will be collected automatically when users log into the application.
Mobile application appreciation (acceptability) | 2-weeks post baseline
  The intervention appreciation will be measured with the User Version of the Mobile Application Rating Scale (uMARS) (Stoyanov, Hides, Kavanagh, & Wilson, 2016). The uMARS is a 20-item measure that includes 4 objective quality subscales regarding engagement, functionality, aesthetics, and information quality and 1 subjective quality subscale. Each item is rated on a 5-point scale ranging from inadequate (+1) to excellent (+5). The possible total score ranges between 20 and 100; a higher scores indicates a higher appreciation.

SECONDARY OUTCOMES:
Online recruitment rate (feasibility of the study processes) | 6 months
  The recruitment rate (ie. number of participants who signed the inform consent form) will be assessed.
Adherence to data collection methods (feasibility of the study processes) | baseline, 4-weeks post baseline, 8-weeks post baseline
  The adherence to data collection methods (ie. number of missing data) will be assessed.
Attrition rate (feasibility of the study processes) | 6 months
  The attrition rate will be measured by taking into account the proportion of participants who completed only the baseline but no follow-up assessment (study dropouts). The proportion of participants who completed the baseline assessment and only one follow-up and the proportion of study completers (who completed all assessments) will also be determined. Loss-to-follow up in both intervention groups will be compared (experimental VS control groups).

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Montréal, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.crsi.umontreal.ca/en/
- See also: Related Info — https://etudejointeffort.ca/home